CLINICAL TRIAL: NCT04256694
Title: Rapid Antigen Test Results for Group A Streptococcus in Healthy Adults
Brief Title: Rapid Strep Test Results
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kendall Healthcare Group, Ltd. (Industry)
Collaborators: Florida International University (Other)
Responsible Party: Sponsor
Other Study IDs: 108360
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Strept Throat
Keywords: Carrier rate; Rapid antigen test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Adult Subjects
  Interventions: Diagnostic Test: Rapid Antigen Test for Group A Streptococcus

INTERVENTIONS:
Diagnostic Test: Rapid Antigen Test for Group A Streptococcus — Rapid strep tests will be performed by throat swab of healthy adult volunteers.

SUMMARY:
This is a prospective study seeks to determine how often a rapid antigens test for group A streptococcus is positive in healthy adults

DETAILED DESCRIPTION:
The Unites States recommends the use of rapid antigen tests, but a number of other countries do not, citing a high prevalence of streptococcal carriers and only moderate sensitivity of rapid antigen tests [1]. Indeed, to fully understand when rapid antigen tests should be used, we need to know the streptococcal carrier rate for adults in the United States. Although there is a fair amount of data in this regard for children [2,3], the only study to report this value for adults was from over 20 years ago and was from Sweden [4]. That studied reported a Group A Streptococcus (GAS) carrier rate of 2.4-3.7% in healthy adults.

Given how many patients seek medical care for sore throats that may potentially be streptococcal pharyngitis, the investigators believe more data about the GAS carrier rate and the rate of false positive rapid antigen tests is necessary. Thus, the investigators propose a prospective study to evaluate the rate of positive rapid antigen tests in healthy adult patients in our community.

The investigators will perform rapid antigen tests for GAS on healthy adult subjects without any symptoms. Consenting patients will fill out a brief data collection form about their medical history, and an investigator will perform a rapid antigen throat swab to assess for GAS. The results of the rapid antigen test will be recorded, and a logistic regression analysis will be performed to determine if certain factors within the subject's medical history are predictive of positive rapid strep tests.

ELIGIBILITY:
Inclusion Criteria:

* Any person at least 18 years old

Exclusion Criteria:

* pregnant
* prisoners
* currently taking antibiotics
* any acute symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers, primarily from subjects known to the investigators.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-02-05 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
% Positive Rapid Antigen Strep Tests | The throat will be swabbed, and the swab will be immediately analyzed. The results are available after five minutes.
  % of positive rapid antigen strep tests amongst all volunteers

SECONDARY OUTCOMES:
Predictors of Positive Strep Tests | After enrollment of all subjects, a logistic regression analysis will be performed.
  Logistic regression analysis will assess if any of the following are significant predictors of positive strep tests: age, gender, race/ethnicity, chronic medical problems, whether or not the patient has had antibiotics within last month, whether or not they have a history of strep throat, and whether or not they are a medical student or healthcare professional.

CONTACTS AND LOCATIONS:
Overall Officials: Tony Zitek, MD, Principal Investigator — Kendall Healthcare Group, Ltd.
Locations (1):
- Kendall Regional Medical Center, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Matthys J, De Meyere M, van Driel ML, De Sutter A. Differences among international pharyngitis guidelines: not just academic. Ann Fam Med. 2007 Sep-Oct;5(5):436-43. doi: 10.1370/afm.741. PMID 17893386
- [Background] Shaikh N, Leonard E, Martin JM. Prevalence of streptococcal pharyngitis and streptococcal carriage in children: a meta-analysis. Pediatrics. 2010 Sep;126(3):e557-64. doi: 10.1542/peds.2009-2648. Epub 2010 Aug 9. PMID 20696723
- [Background] Oliver J, Malliya Wadu E, Pierse N, Moreland NJ, Williamson DA, Baker MG. Group A Streptococcus pharyngitis and pharyngeal carriage: A meta-analysis. PLoS Negl Trop Dis. 2018 Mar 19;12(3):e0006335. doi: 10.1371/journal.pntd.0006335. eCollection 2018 Mar. PMID 29554121
- [Background] Gunnarsson RK, Holm SE, Soderstrom M. The prevalence of beta-haemolytic streptococci in throat specimens from healthy children and adults. Implications for the clinical value of throat cultures. Scand J Prim Health Care. 1997 Sep;15(3):149-55. doi: 10.3109/02813439709018506. PMID 9323783